CLINICAL TRIAL: NCT05513248
Title: Perioperative Outcomes of Anatomic Lung Resections in Patients Who Recovered From Coronavirus Disease 2019 (COVID-19): a Two-Year Retrospective Case Series
Brief Title: Perioperative Outcomes of Anatomic Lung Resections in Patients Who Recovered From Coronavirus Disease 2019
Status: Completed | Type: Observational
Sponsor: Lung Center of the Philippines (Other)
Responsible Party: Principal Investigator, Alexander H. Tuliao, Medical Officer III, Lung Center of the Philippines
Other Study IDs: LCP-SF-013-2022
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: COVID-19; Lung Cancer; Lung TB; Hemoptysis
MeSH Terms: conditions — COVID-19; Lung Neoplasms; Tuberculosis, Pulmonary; Hemoptysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who recovered from COVID-19: patients with previous COVID-19 infection who underwent anatomic lung resection (segmentectomy, lobectomy, bilobectomy or pneumonectomy)
  Interventions: Procedure: anatomic lung resection

INTERVENTIONS:
Procedure: anatomic lung resection — includes minimally invasive or open lung segmentectomy, lobectomy, bilobectomy and pneumonectomy

SUMMARY:
This study will determine the outcomes of anatomic lung resections in patients who recovered from coronavirus disease 2019 (COVID-19) disease by describing the morbidity and mortality as well as the length of postoperative hospital stay.

DETAILED DESCRIPTION:
This study will be conducted at the Lung Center of the Philippines. The study design is a retrospective case series implemented via chart review. Online and written patient records will be reviewed to determine the baseline patient characteristics and the preoperative outcomes. Patients who recovered from COVID-19 will be selected from those who underwent anatomic lung resection from June 1, 2020 to May 31, 2022. This study will be done in accordance with the Helsinky Declaration and Good Clinical Practice Guidelines, and will be subject for approval of the institutional Ethics and Technical Review Boards. Descriptive statistics will be used to describe patient characteristics and perioperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* underwent anatomic lung resection
* previous COVID-19 infection documented by nasopharyngeal swab RT-PCR or GeneXpert
* with negative nasopharyngeal swab RT-PCR or GeneXpert prior to lung resection

Exclusion Criteria:

* with incomplete patient records

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who recovered from COVID-19, and who underwent anatomic lung resection (segmentectomy, lobectomy, bilobectomy or pneumonectomy)
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Mortality rate | perioperative period (up to 30 days after anatomic lung resection)
  proportion of patients who died due to perioperative complications
Major complication rate | perioperative period (up to 30 days after anatomic lung resection)
  proportion of patients who develop acute kidney injury, acute myocardial infarction, acute respiratory distress syndrome (ARDS), acute respiratory failure, atelectasis requiring intervention, bronchopleural fistula, empyema thoracis, hemothorax, pneumonia, stroke or venous thromboembolism
Minor complication rate | perioperative period (within 30 days after anatomic lung resection)
  proportion of patients who develop atrial fibrillation, pneumothorax or prolonged air leak
Length of postoperative hospital stay | perioperative period (up to 30 days after anatomic lung resection)
  time duration from surgery to discharge order

CONTACTS AND LOCATIONS:
Overall Officials: Alexander H Tuliao, MD, Principal Investigator — Lung Center of the Philippines
Locations (1):
- Lung Center of the Philippines, Quezon City, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Patient baseline characteristics and outcomes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5 years

REFERENCES:
- [Background] Sakai T, Azuma Y, Aoki K, Wakayama M, Miyoshi S, Kishi K, Tateda K, Homma S, Iyoda A. Elective lung resection after treatment for COVID-19 pneumonia. Gen Thorac Cardiovasc Surg. 2021 Jul;69(7):1159-1162. doi: 10.1007/s11748-021-01630-4. Epub 2021 Apr 3. PMID 33811611
- [Background] Testori A, Perroni G, Voulaz E, Crepaldi A, Alloisio M. Pulmonary Lobectomy After COVID-19. Ann Thorac Surg. 2021 Mar;111(3):e181-e182. doi: 10.1016/j.athoracsur.2020.08.004. Epub 2020 Sep 25. PMID 32987024
- [Background] Nefedov A, Mortada M, Novitskaya T, Patsyuk A, Kozak A, Yablonskii P. Lobectomy with pathological examination in lung cancer patients who recovered from COVID-19. Gen Thorac Cardiovasc Surg. 2021 Aug;69(8):1258-1260. doi: 10.1007/s11748-021-01632-2. Epub 2021 Apr 9. PMID 33837476
- [Background] Diaz A, Bujnowski D, McMullen P, Lysandrou M, Ananthanarayanan V, Husain AN, Freeman R, Vigneswaran WT, Ferguson MK, Donington JS, Madariaga MLL, Abdelsattar ZM. Pulmonary Parenchymal Changes in COVID-19 Survivors. Ann Thorac Surg. 2022 Jul;114(1):301-310. doi: 10.1016/j.athoracsur.2021.06.076. Epub 2021 Jul 31. PMID 34343471
- [Background] COVIDSurg Collaborative; GlobalSurg Collaborative. Timing of surgery following SARS-CoV-2 infection: an international prospective cohort study. Anaesthesia. 2021 Jun;76(6):748-758. doi: 10.1111/anae.15458. Epub 2021 Mar 9. PMID 33690889